CLINICAL TRIAL: NCT00148694
Title: A Phase II Trial of Cisplatin in Early Stage ER-, PR-, HER-2 Negative Breast Cancer
Brief Title: Preoperative Cisplatin in Early Stage Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other); Brigham and Women's Hospital (Other); Breast Cancer Research Foundation (Other)
Responsible Party: Principal Investigator, Judy E. Garber, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-183
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer
Keywords: Cisplatin; Early Stage Breast Cancer; ER Negative Breast Cancer; PR Negative Breast Cancer; HER-2 Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention single arm (Experimental): Cisplatin 75mg/m2 q21 days x 4 pre-surgery
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Cisplatin — Intravenously once every three weeks for a total of 12 weeks

SUMMARY:
The purpose of this study is to find out what effects the preoperative therapy cisplatin will have on patients with early stage estrogen receptor-negative (ER-), progesterone receptor-negative (PR-), or HER-2 negative breast cancer.

DETAILED DESCRIPTION:
Before starting treatment patients will undergo placement of a clip into the tumor bed so the surgeon can locate the site of the tumor at the time of surgery.

Patients will receive cisplatin intravenously once every three weeks for a total of 4 cycles or 12 weeks of treatment.

After completion of cisplatin, patients will undergo surgery to remove any tumor that remains and to assess the tissue to see if tumor cells remain in the breast.

Patients may receive a second breast MRI and biopsy 7-14 days after treatment begins to see whether we can identify tumors that will ultimately respond to cisplatin with a rapid evaluation.

Patients will receive study treatment for approximately 12 weeks unless unacceptable toxicity occurs. After surgery patients will receive standard adjuvant therapy based on discussion with their physician. Follow-up progress will occur for several years.

ELIGIBILITY:
Inclusion Criteria:

* All tumors must be ER-, PR- and HER-2 negative.
* Age > 18 years
* ECOG performance status of less than or equal to 1
* Absolute neutrophil count (ANC) > 1,500/mm3
* Hemoglobin > 9mm/dl
* Platelets > 100,000/mm3
* Creatinine < 1.5mg/dl
* Glucose < 200mg/dl
* Bilirubin < 1.5 x upper limit of normal (ULN)
* SGOT < 3.0 x ULN

Exclusion Criteria:

* Prior chemotherapy treatment
* Pregnant or breast-feeding women
* History of serious illness, medical or psychiatric condition requiring medical management
* Uncontrolled infection
* Renal dysfunction
* Active or severe cardiovascular or pulmonary disease
* Peripheral neuropathy of any etiology that exceeds grade 1
* Prior history of malignancy
* Uncontrolled diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2004-07; Primary Completion 2006-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To determine the clinical response after preoperative therapy with cisplatin in ER-, PR-, HER-2 negative early breast cancer patients

SECONDARY OUTCOMES:
To determine the pathologic complete response after preoperative therapy with cisplatin in this patient population

CONTACTS AND LOCATIONS:
Overall Officials: Judy E. Garber, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Silver DP, Richardson AL, Eklund AC, Wang ZC, Szallasi Z, Li Q, Juul N, Leong CO, Calogrias D, Buraimoh A, Fatima A, Gelman RS, Ryan PD, Tung NM, De Nicolo A, Ganesan S, Miron A, Colin C, Sgroi DC, Ellisen LW, Winer EP, Garber JE. Efficacy of neoadjuvant Cisplatin in triple-negative breast cancer. J Clin Oncol. 2010 Mar 1;28(7):1145-53. doi: 10.1200/JCO.2009.22.4725. Epub 2010 Jan 25. PMID 20100965
- [Result] Birkbak NJ, Wang ZC, Kim JY, Eklund AC, Li Q, Tian R, Bowman-Colin C, Li Y, Greene-Colozzi A, Iglehart JD, Tung N, Ryan PD, Garber JE, Silver DP, Szallasi Z, Richardson AL. Telomeric allelic imbalance indicates defective DNA repair and sensitivity to DNA-damaging agents. Cancer Discov. 2012 Apr;2(4):366-375. doi: 10.1158/2159-8290.CD-11-0206. Epub 2012 Mar 22. PMID 22576213